CLINICAL TRIAL: NCT04757428
Title: Clinical Evaluation of Lithium Disilicate and Hybrid Nano-ceramic Anterior Endocrowns (Randomized Clinical Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Abou-steit, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD 37/7/22
Record Dates: First submitted 2021-01-31; First posted 2021-02-17 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Personal Satisfaction
Keywords: Lithium disilicate; hybrid ceramic
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lithium disilicate (Active Comparator): The intervention will be: Prosthetic endocrown
  Interventions: Procedure: Endocrown
- Hybrid nanoceramic (Active Comparator): The intervention will be: Prosthetic endocrown
  Interventions: Procedure: Endocrown

INTERVENTIONS:
Procedure: Endocrown — Endocrown

SUMMARY:
the aim of this study was to evaluate the clinical performance of two CAD/CAM materials, hybrid nano-ceramic and lithium disilicate ceramic, in the fabrication of anterior endocrowns in patients with anterior endodontically treated teeth. While the postulated null hypothesis of this study was that there will be no significant difference between the performance of hybrid nanoceramic and lithium disilicate anterior endocrowns in patients with endodontically treated teeth.

ELIGIBILITY:
Inclusion Criteria:

* Patients with good oral hygiene
* Patients having one or more endodontically treated molars that need prosthetic restoration.
* Molars should have enough tooth structure for endocrown restoration with minimum 3 walls with thickness not less than 1.5 mm and gingival step placed supragingival
* Fully erupted molars
* Molars free of developmental defect
* Healthy periodontium
* Absence of periapical pathosis
* Acceptable endodontic treatment and proper bone support

Exclusion Criteria:

* Patients with bad oral hygiene
* Patients with active periodontal disease
* Patients with missing teeth opposing to the area intended for restoration
* Patients with parafunctional habits or psychiatric problems or unrealistic expectation.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 2 years
  Using Binary Visual Analogue scale (Satisfied/ not satisfied)

SECONDARY OUTCOMES:
Shade matching | 2 years
  Using the modified United States Public Health Service criteria (Modified USPHS)- categorical

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Sh Abou-steit, PhD, Principal Investigator — Lecturer of Fixed Prosthodontics
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] da Cunha LF, Gonzaga CC, Pissaia JF, Correr GM. Lithium silicate endocrown fabricated with a CAD-CAM system: A functional and esthetic protocol. J Prosthet Dent. 2017 Aug;118(2):131-134. doi: 10.1016/j.prosdent.2016.10.006. Epub 2017 Jan 13. PMID 28089332
- [Background] Wang F, Yu T, Chen J. Biaxial flexural strength and translucent characteristics of dental lithium disilicate glass ceramics with different translucencies. J Prosthodont Res. 2020 Jan;64(1):71-77. doi: 10.1016/j.jpor.2019.04.007. Epub 2019 May 11. PMID 31088735
- [Background] Rosentritt M, Preis V, Behr M, Hahnel S. Influence of preparation, fitting, and cementation on the vitro performance and fracture resistance of CAD/CAM crowns. J Dent. 2017 Oct;65:70-75. doi: 10.1016/j.jdent.2017.07.006. Epub 2017 Jul 19. PMID 28734997
- [Background] Tribst JPM, Dal Piva AMO, Madruga CFL, Valera MC, Borges ALS, Bresciani E, de Melo RM. Endocrown restorations: Influence of dental remnant and restorative material on stress distribution. Dent Mater. 2018 Oct;34(10):1466-1473. doi: 10.1016/j.dental.2018.06.012. Epub 2018 Jun 21. PMID 29935769
- [Background] da Fonseca GF, Dal Piva AM, Tribst JP, Borges AL. Influence of Restoration Height and Masticatory Load Orientation on Ceramic Endocrowns. J Contemp Dent Pract. 2018 Sep 1;19(9):1052-1057. PMID 30287703
- [Background] Schaefer O, Watts DC, Sigusch BW, Kuepper H, Guentsch A. Marginal and internal fit of pressed lithium disilicate partial crowns in vitro: a three-dimensional analysis of accuracy and reproducibility. Dent Mater. 2012 Mar;28(3):320-6. doi: 10.1016/j.dental.2011.12.008. Epub 2012 Jan 21. PMID 22265824
- [Background] Shamseddine L, Mortada R, Rifai K, Chidiac JJ. Marginal and internal fit of pressed ceramic crowns made from conventional and computer-aided design and computer-aided manufacturing wax patterns: An in vitro comparison. J Prosthet Dent. 2016 Aug;116(2):242-8. doi: 10.1016/j.prosdent.2015.12.005. Epub 2016 Mar 3. PMID 26948080
- [Background] Belleflamme MM, Geerts SO, Louwette MM, Grenade CF, Vanheusden AJ, Mainjot AK. No post-no core approach to restore severely damaged posterior teeth: An up to 10-year retrospective study of documented endocrown cases. J Dent. 2017 Aug;63:1-7. doi: 10.1016/j.jdent.2017.04.009. Epub 2017 Apr 27. PMID 28456557
- [Background] Tzimas K, Tsiafitsa M, Gerasimou P, Tsitrou E. Endocrown restorations for extensively damaged posterior teeth: clinical performance of three cases. Restor Dent Endod. 2018 Aug 22;43(4):e38. doi: 10.5395/rde.2018.43.e38. eCollection 2018 Nov. PMID 30483462
- [Background] Sedrez-Porto JA, Rosa WL, da Silva AF, Munchow EA, Pereira-Cenci T. Endocrown restorations: A systematic review and meta-analysis. J Dent. 2016 Sep;52:8-14. doi: 10.1016/j.jdent.2016.07.005. Epub 2016 Jul 12. PMID 27421989
- [Background] Furtado de Mendonca A, Shahmoradi M, Gouvea CVD, De Souza GM, Ellakwa A. Microstructural and Mechanical Characterization of CAD/CAM Materials for Monolithic Dental Restorations. J Prosthodont. 2019 Feb;28(2):e587-e594. doi: 10.1111/jopr.12964. Epub 2018 Aug 18. PMID 30121945
- [Background] Otto T, Mormann WH. Clinical performance of chairside CAD/CAM feldspathic ceramic posterior shoulder crowns and endocrowns up to 12 years. Int J Comput Dent. 2015;18(2):147-61. English, German. PMID 26110927